CLINICAL TRIAL: NCT02784834
Title: Phase I Clinical Trial to Evaluate Dimethylfumarate (DMF) in Relapsed/Refractory Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma.
Brief Title: Dimethylfumarate (DMF) in Relapsed/Refractory CLL/SLL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Michael Choi (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor-Investigator, Michael Choi, Associate Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 151657
Record Dates: First submitted 2016-05-23; First posted 2016-05-27 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL; cancer; DMF; SLL; dimethylfumarate; relapsed; refractory
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Recurrence | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dimethyl fumarate (DMF) (Experimental): Cohort 1: dimethyl fumarate 120 mg PO BID (approximately 12 hours apart) for 2 x 28 day cycles.
  Cohort 2: dimethyl fumarate 120 mg PO BID (approximately 12 hours apart) for 1 week, then escalating to the assigned dose of (240mg PO BID for the remainder of 2 x 28 day cycles.
  Cohort 3: dimethyl fumarate 120 mg PO BID for 1 week, then escalate to the dose of 360mg PO BID for the remainder of 2 x 28 day cycles.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate
  Other Names: Tecfidera; DMF

SUMMARY:
The purpose of the study is to investigate the safety of the investigational drug called dimethylfumarate (DMF). DMF is a type of drug called an immunomodulatory drug. This drug is approved by the United States (U.S.) Food and Drug Administration (FDA) as a treatment for patient with multiple sclerosis.

Although there is evidence from tests on laboratory animals that DMF can decrease the number of CLL cells, we do not know if this will work in humans with CLL. This drug will be given to humans with CLL for the first time in this study. Therefore, the goal of this study is to see if DMF is safe and tolerable in study participants. Participants will be evaluated to find out what effects (good and bad) DMF has on the body and see how long the drug stays in the body.

DETAILED DESCRIPTION:
This is a phase I clinical trial to evaluate the safety, tolerability, and maximum tolerated dose of DMF in patients with chronic lymphocytic leukemia. Patients with relapsed/refractory CLL not amenable to available therapies are eligible. This patient population is in need of novel therapies, particularly if progressing after, intolerant of, or unable to receive oral tyrosine kinase inhibitors (ie ibrutinib, idelalisib).

For Dose Level 1, DMF (Tecfidera formulation) will be administered at a dose of 120 mg PO BID (approximately 12 hours apart) for 2 x 28 day cycles.

For Dose Level 2, DMF will be administered at the currently used dose for patients with multiple sclerosis: at the standard FDA approved dose of 120 mg PO BID (approximately 12 hours apart) for 1 week, then escalating to the assigned dose of (240mg PO BID for the remainder of 2 x 28 day cycles. The 1 week lead-in at 120 mg is to assist in toleration and initial side effects and is as per the standard prescribing information.

For Dose Level 3, DMF will be administered at the currently used dose for patients with multiple sclerosis: 120 mg PO BID for 1 week, then escalate to the dose of 360mg PO BID for the remainder of 2 x 28 day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and phenotypic verification of B cell CLL/ SLL/ or MBL and measurable disease.
* Relapsed or refractory disease
* Previously treated with at least 1 regimen for CLL/SLL
* Not appropriate or amenable to all approved therapies.

  * All patients must have progressed on or after B-cell receptor targeted kinase inhibitor (eg: ibrutinib, idelalisib, ACP-196, CC-292), unless there is a relative contraindication (eg: history of recent bleeding, history of atrial fibrillation, unacceptable high out-of-pocket cost despite patient assistance programs).
  * Patients with Del(17p) CLL must have progressed on or after BCL-2 inhibitor therapy (eg: venetoclax), unless there is a relative contraindication (eg: Creatinine clearance < 50ml/min, or unable to monitor for TLS due to living remotely from the medical center, unacceptably high out-of-pocket cost).
  * Patients must have received a CD20-directed monoclonal antibody (eg: obinutuzumab, ofatumumab, rituximab), unless there is a relative contraindication (eg: history of hepatitis virus infection).
* Has recovered from the toxic effects of prior therapy to their clinical baseline.
* Women of childbearing potential must agree not to become pregnant for the duration of the study.
* Both men and women must agree to use a barrier method of contraception for the duration of the study and until 8 weeks after the final dose.
* Subjects must have at least one of the following indications for treatment:

  * Symptomatic or progressive splenomegaly;
  * Symptomatic lymph nodes, nodal clusters, or progressive lymphadenopathy;
  * Progressive anemia;
  * Progressive thrombocytopenia;
  * Weight loss > 10% body weight over the preceding 6 month period;
  * Fatigue attributable to CLL;
  * Fever or night sweats for > 2 weeks without evidence of infection;
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period or an anticipated doubling time of less than 12 months.
* ECOG performance status of 0-2.
* Adequate hematologic function
* Adequate renal function
* Adequate hepatic function

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study.
* Patients who are currently receiving another investigational agent are excluded.
* Patients who have had chemotherapy (e.g., purine analogues, alkylating agents), radiation therapy, or participation in any investigational drug treatment within 4 weeks of initiation of DMF or at any time during the study.
* Patients who have had prior (within 8 weeks of initiation of DMF) or concurrent antibody therapy directed against CLL (i.e. Rituxan and Campath)
* Patients who have had tyrosine kinase inhibitor therapy (eg: ibrutinib or idelalisib) within 7 half lives (or 28 days, which ever is shorter) of initiation of DMF.
* Current infection requiring parenteral antibiotics.
* Active malignancy within the previous 2 years (other than completely resected non-melanoma skin cancer or carcinoma in situ).
* Insufficient recovery from surgical-related trauma or wound healing.
* Impaired cardiac function including any of the following:

  * Myocardial infarction within 6 months of starting study drug;
  * Other clinically significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Choi, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dimethyl Fumarate (DMF): Cohort 1: dimethyl fumarate 120 mg PO BID (approximately 12 hours apart) for 2 x 28 day cycles.
Period: Overall Study
Arm/Group | Dimethyl Fumarate (DMF)
Started | 2
Completed | 1
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicity
Description: The incidence of dose limiting toxicities (DLTs) will be used to define the maximum tolerated dose or biologically active dose for potential phase 2 studies.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Dimethyl Fumarate (DMF)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dimethyl Fumarate (DMF) (N=2)
Allergic Reaction (Immune system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Thrombocytopenia (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT02784834/Prot_SAP_000.pdf